CLINICAL TRIAL: NCT03987542
Title: Outcome Following Truncation of Asparaginase in the NOPHO ALL2008 Protocol
Brief Title: Outcome Following Truncation of Asparaginase
Status: Completed | Type: Observational
Sponsor: Birgitte Klug Albertsen (Other)
Responsible Party: Sponsor-Investigator, Birgitte Klug Albertsen, M.D., PhD, Associate Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: Asparaginase_truncation_NOPHO
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Relapse Leukemia
Keywords: Acute lymphoblastic leukemia; Asparaginase; Truncation; Toxicitities
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Patients who had their asparaginase treatment truncated or had no asparaginase enzyme activity.
- Unexposed: Patients who did not have their asparaginase treatment truncated and had measurable asparaginase enzyme activity

SUMMARY:
This study aimed to investigate the outcome of patients who had their asparaginase treatment truncated in the NOPHO ALL2008 protocol.

DETAILED DESCRIPTION:
Overall survival for children with ALL is now above 90% in several protocols, but asparaginase associated toxicities still constitutes a significant problem as they, besides causing acute morbidity and mortality, can cause truncation of treatment with a subsequent increased risk of relapse.

The most frequent toxicities causing asparaginase truncations are hypersensitivity, pancreatitis and thrombosis. Especially hypersensitivity constitutes a problem due to silencing antibodies, not only in patients with clinical hypersensitivity but also in patients without clinical symptoms (silent inactivation).

In the NOPHO ALL2008 protocol asparaginase associated toxicities and truncation of asparaginase have been registered since the protocol opened in 2008. In addition asparaginase enzyme activity measurements have been done before every asparaginase administration and analyzed retrospectively.

The primary aim of this study was to investigate if patients with truncation of asparaginase or lack of asparaginase enzyme activity had a different risk of relapse compared to patients who received full asparaginase treatment. Secondary we aimed to explore if patients who received less than 50% of their planned asparaginase dosages had a different risk of relapse compared to those who received 50% or more.

ELIGIBILITY:
Inclusion Criteria:

- Children treated according to the NOPHO ALL2008 protocol from the 1st of July 2008 - 28th of February 2016.

Exclusion Criteria:

* Bilineage ALL
* Pre-treatment with glucocorticosteroids or other antileukemic agents for more than 1 week
* ALL predisposition syndromes
* Previous cancer
* Off protocol administration of additional chemotherapy during induction therapy
* Sexually active females not using contraception

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 1-17.9 years at time of diagnosis.
Sampling Method: Probability Sample
Enrollment: 1401 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Risk of relapse | 5 years
  Do patients with truncation of asparaginase treatment or no enzyme activity (truncated) have a different risk of relapse compared to patients who have not been truncated and who have measurable enzyme activity (non-truncated)

SECONDARY OUTCOMES:
50% of asparagine doses | 5 years
  Do patients who receive less than 50% of their planned asparaginase dosages have a different risk of relapse compared to those who receive 50% or more.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Pediatrics Skejby Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gottschalk Hojfeldt S, Grell K, Abrahamsson J, Lund B, Vettenranta K, Jonsson OG, Frandsen TL, Wolthers BO, Marquart HV, Vaitkeviciene G, Lepik K, Heyman M, Schmiegelow K, Albertsen BK. Relapse risk following truncation of pegylated asparaginase in childhood acute lymphoblastic leukemia. Blood. 2021 Apr 29;137(17):2373-2382. doi: 10.1182/blood.2020006583. PMID 33150360